CLINICAL TRIAL: NCT06486922
Title: Starting Early to Prevent Obesity Using Telehealth (StEP OUT): Intervention Development Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Michelle Katzow, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-1078 Aim 2
Record Dates: First submitted 2024-06-20; First posted 2024-07-05 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Child Obesity; Breast Feeding; Feeding Behavior; Nutrition, Healthy
MeSH Terms: conditions — Pediatric Obesity; Breast Feeding; Feeding Behavior

STUDY DESIGN:
Intervention Model Description: Sequential, single arm, intervention development study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- StEP OUT Intervention (Experimental): See intervention description
  Interventions: Behavioral: StEP OUT

INTERVENTIONS:
Behavioral: StEP OUT — The details of program structure and content will evolve as the study progresses based on feedback from participants, interventionists, and the community advisory board. Initially, we will plan to have 5 formal sessions structured as groups with multiple participants receiving the session simultaneously, primarily via remote videoconference, though sessions may occur individually, based on participant schedule and preference. All sessions are designed to be supportive, educational, and interactive, with opportunities to practice skills and discuss feeding and parenting concerns.

SUMMARY:
The goal of this intervention development study is to optimize the Starting Early to Prevent Obesity Using Telehealth (StEP OUT) intervention for feasibility and acceptability, using human-centered design and community-engaged research methods.

DETAILED DESCRIPTION:
This intervention development study will enroll three to four consecutive cohorts to receive Starting Early to Prevent Obesity Using Telehealth (StEP OUT), an online, group-based nutrition education and parenting support program beginning in the third trimester of pregnancy and continuing through the first four to six months of infancy. It is tailored to Hispanic/Latinx families. StEP OUT will be delivered by a registered dietician/certified lactation counselor in coordination with the Long Island Jewish Medical Center Special Supplemental Nutrition Program for Women, Infants, and Children (LIJ WIC). The StEP OUT curriculum is based on the Starting Early Program (StEP), which uses didactic instruction, reflective discussion, interactive demonstrations, and hands-on practicing of skills to support prenatal nutrition and healthy early infant feeding practices. The details of program structure and content will evolve as the study progresses based on feedback from participants, interventionists, and our Community Advisory Board. Initially, we will plan to have 5 formal sessions structured as groups with multiple participants receiving the session simultaneously, primarily via remote videoconference, though sessions may occur individually, based on participant schedule and preference. Each session will conclude with a structured feedback discussion designed to elicit targets and strategies for further program adaptation. We will collect feasibility and acceptability data after each session and at the end of the five-session program for each cohort. The iterative intervention adaptation process will be complete once all participants rate the intervention as "acceptable" or higher and fidelity is 90% or higher. We anticipate meeting this benchmark after 3 cohorts but may need to recruit an additional cohort to test subsequent adaptations, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant with at least 14 weeks estimated gestational age
* Self-identify as Hispanic/Latinx
* Speak fluent English or Spanish
* At least 18 years of age
* Has a phone or device to participate in video calls
* Receiving or eligible to receive WIC benefits

Exclusion Criteria:

* Diminished mental capacity
* Serious medical or psychiatric illness
* Serious fetal illness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-06-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Acceptability | From enrollment through the end of the study after child age 4 months.
  We will use the Sekhon acceptability framework to assess affective attitude, burden, opportunity cost, perceived effectiveness, coherence, ethicality, self-efficacy and general acceptability.
Feasibility | From enrollment to study completion after infant age 4 months.
  Feasibility assessment will include measures of recruitment (number enrolled of those eligible), retention (number who attend all scheduled sessions of those enrolled), fidelity (number of curriculun components delivered of those planned), and attendance (1. Attendance rate: number of participants who attend each sessions of those scheduled to attend; 2. Program dose: number of sessions attended for each participant)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle W Katzow, MD, MS, Principal Investigator — Northwell Health
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No